CLINICAL TRIAL: NCT05973916
Title: A Comprehensive Intervention to Improve the Level of Cleaning and Disinfection of Patients' Units, in Order to Reduce New Acquisitions and Environmental Contamination by Multidrug Resistant Organisms: a Prospective Controlled Crossover Trial, Using VYV Led Lights and Continuous Air Filtering of Patients' Rooms, Coupled With Establishment of a "Patient's Unit Commando" Cleaning Team.
Brief Title: Comprehensive Intervention to Improve Environmental Disinfection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Dror MarChaim, MD, Head of the Unit of Infection Control & Prevention, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 172-22-ASF
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Hospital Acquired Condition
MeSH Terms: conditions — Iatrogenic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive intervention (Experimental): Cleaning of patients' rooms will be subjected to a comprehensive intervention, consisting of: 1) a "patient's unit commando" team for daily and for terminal cleaning, 2) all lights in patients' room are VYV led lights, and 3) in each room, a QleanAir Scandinavia® filtering machine will be placed.
  Interventions: Other: Comprehensive intervention
- Common Practice (No Intervention): Patients' rooms will be cleaned and disinfected according to the current "common practice" as detailed below.

INTERVENTIONS:
Other: Comprehensive intervention — cleaning of patients' rooms will be subjected to a comprehensive intervention, consisting of: 1) a "patient's unit commando" team for daily and for terminal cleaning, 2) all lights in patients' room are VYV led lights, and 3) in each room, a QleanAir Scandinavia® filtering machine will be placed.
  Other Names: VYV led lights; Patient's unit commando; QleanAir Scandinavia® filtering machine
  Arms: Comprehensive intervention

SUMMARY:
A comprehensive intervention to improve the level of cleaning and disinfection of patients' units, in order to reduce new acquisitions and environmental contamination by multidrug resistant organisms: a prospective controlled crossover trial, using VYV led lights and continuous air filtering of patients' rooms, coupled with establishment of a "patient's unit commando" cleaning team.

DETAILED DESCRIPTION:
Background and introduction

As declared by the World Health Organization (WHO) in 2016, antimicrobial resistance among the commonest human pathogens, i.e., the multidrug resistant organisms (MDRO), pose one of the biggest challenges in modern Medicine and one of the biggest threats to humanity. MDROs are prevalent in acute-care hospitals, and in addition are continuously emerging at non-acute-care healthcare settings, and even in the community. The current global SARS-CoV-2 pandemic, further amplifies the enormous burdens imposed by MDROs on hospitalized previously non-sick individuals. The commonest Gram-positive MDROs are methicillin-resistant Staphylococcus aureus (MRSA), vancomycin-resistant enterococci (VRE), and Clostridioides difficile (C. diff). The commonest Gram-negative MDROs are carbapenem-resistant and/or carbapenemase-producing Enterobacterales (CRE), Acinetobacter baumannii (CRAB), and Pseudomonas aeruginosa (CRPA). Acquisition of an MDRO in the hospital is associated with devastating outcomes to the individual patient and with enormous fiscal burden imposed on health facilities. Moreover, In Israel and in many other countries, there are mandatory reporting regulations for certain MDROs, and the rates of MDRO acquisitions serve as "pay per performance" initiatives. This adds additional burden in terms of potential bad reputation and reductions in reimbursements.

The patient's immediate environment, specifically "high-touch surfaces" (e.g., touch screens, monitor, respirator, feeding device, infusion pump, the entire bed, cabin, nurse's call-on button, light switches, fluid balance charts hanged on bed, linen, armchairs, curtains, and so on), serves as reservoir and vector for MDRO distribution and transmission from patient to patient. Therefore, health facilities have strong motivation to improve the level of cleaning and disinfection of patients' immediate environment, in an effort to improve patient safety, quality of clinical care, and reduce hospital costs while improving its reputation.

Many items commonly used in traditional and routine care of hospitalized patients, have been described as reservoirs and/or fomites for transmission of pathogens, which can lead to nosocomial MDRO-related outbreaks. Environmental remnants of MDROs on immediate high touch surfaces spread from patient to patient through staff, shared equipment, or directly from patient to patient (less common). While a carrier of a specific MDRO reside in his/her room or unit, the same MDRO can be isolated (frequently in high inoculums) from the patient's immediate environment (e.g. bedrail, monitor, infusion pump), from high-touch surfaces (e.g., light switches, water taps, nurse's call-on button), and even from distant locations in the room (e.g. ceiling). MDROs can remain viable and survive in those transmitting-prone environmental locations for prolonged periods, long after the previous carrier who contaminated the environment had been discharged.

The levels of environmental cleaning and disinfection of high-touch surfaces, is known to be low in hospitals. The current cleaning guidelines at Shamir Medical Center (SMC), as per the Israeli MOH regulations, are as follows: while the patient is in their bed, the unit is subjected to daily cleaning, and after the patient leaves, the unit is subjected to "terminal cleaning", a supposable standardized enhanced cleaning protocol. Recurrent audits and observations from all over the world clearly suggests that the level of cleaning and disinfection of patients' environments in acute-care hospitals is unsatisfactory most hours of the day. In order to improve this crucial aspect associated with MDRO transmission and spread in hospitals, a multidisciplinary approach is warranted, with implementation of novel solutions both technological, and with regards to aspects associated with human capital. To add an additional complexity to the situation, in Israeli hospitals, as in many other countries, the responsibility of cleaning/disinfecting patient's immediate environment, is divided. The bed, bedside table, infusion pump, monitor, cables and additional immediate surroundings of an individual patient, are cleaned by nurse assistants, while the floor, sink, toilets, light switches and walls (shared by all room occupants), are cleaned by environmental services (EVS) personnel. This separation in responsibilities creates eventual gaps in the overall level of cleaning/disinfection of certain items, which are frequently associated with MDRO transmission. There are continuous shortages both in terms of full time effort (fte) allocation, and in terms of specified professional training, among these two frequently neglected sectors (i.e., nurse assistants and EVS personnel). The employment turnaround time of these personnel sectors is very high, with no establishment of a stable local base of knowledge and expertise. In order for an intervention that improves the level of cleaning /disinfection of patients' environment to be successful, human capital considerations must be acknowledged and addressed. A designated team (referred to as "cleaning commando" in certain facilities), responsible to all the various aspects associated with cleaning and disinfecting the patient's environment, but have no other additional responsibilities, and is managed by the same management, could theoretically improve the human capital aspects associated with improving the level of cleaning/disinfecting patients' environments in hospitals.

The market is flooded in recent years, and even more since the emergence of the SARS-CoV-2 pandemia, with novel technologies that aim to improve the level of environmental disinfection of patients' surroundings and high-touch surfaces. These technologies should always be applied on top of an effective process of cleaning, which is always executed by humans. These technologies only add an additional level of mechanized controlled process for enhancing environmental disinfection, but could never replace the necessity of an established effective and monitored process of initial cleaning, a process that should be executed, as mentioned above, by trained and centrally managed personnel. Initially, many of the technologies in this field of immediate environment disinfection, were applied on empty patients' units only. This creates many operational complexities in busy acute-care hospitals, with fast turnaround time of hospitalized beds. The "new generation" of technologies, are aimed to disinfect patients' immediate environment, continuously, while the patients reside in the unit. On the one hand, technology needs to be effective and bactericidal, but on the other hand, concentrations of the active disinfecting ingredients or materials, should not be toxic and endanger patients under no circumstances. Continuously disinfecting surfaces by using VYV led lights, and filtering the air by using the QleanAir Scandinavia® device, are both licensed to operate while the patients are in the room. Both are "effective" in-vitro against the six groups of MDROs mentioned above. This could theoretically add an additional mode for prevention of MDRO transmission and spread in hospitals. However, controlled clinical data, with 'real' clinical outcomes, pertaining to the actual efficacy of these technologies in preventing MDRO acquisitions, are absent. In order to convince stakeholder administrators to invest in implementation of certain preventing technologies, clinical studies, analyzing the effectiveness of technologies in preventing actual clinical outcomes, are warranted.

Crossover design is considered today the gold standard methodology in the clinical research field of infection control and hospital epidemiology. This design enables to control for multiple confounders, associated with the Hawthorne effect, which is very common in studies assessing the controlled efficacy of a certain infection control newly implemented intervention.

In order to reduce the environmental contamination by MDRO carriers, and the incidence of MDRO acquisitions in hospitals by naïve patients, we aim to implement a comprehensive and multifactorial intervention, to improve the level of cleaning/disinfecting patients' immediate environment. The suggested intervention will contain components associated with human capital and with the implementation of two advanced technologies. We aim to trial this comprehensive intervention, in a prospective crossover design, in a 'real-world' clinical scenario, analyzing its efficacy on 'hard' and direct clinical outcomes.

Study hypotheses

1. A comprehensive intervention (consisting of establishing a "patient's unit commando" team, while continuously disinfecting patient's unit by using VYV led lights and QleanAir Scandinavia® air filtering device) will reduce the rate of new carriage acquisitions of the MDROs: 1) MRSA, 2) VRE, 3) CRE, 4) A. baumannii, 5) P. aeruginosa, and 6) C. difficile.
2. A comprehensive intervention (consisting of establishing a "patient's unit commando" team, while continuously disinfecting patient's unit by using VYV led lights and QleanAir Scandinavia® air filtering device) will reduce the incidence of hospital-acquired bloodstream infections (HA-BSI).
3. A comprehensive intervention (consisting of establishing a "patient's unit commando" team, while continuously disinfecting patient's unit by using VYV led lights and QleanAir Scandinavia® air filtering device) will reduce the incidence of hospital-acquired urinary-tract infections (HAUTI).

   Study Aim
   1. Analyze the role of a comprehensive intervention (consisting of establishing a "patient's unit commando" team, while continuously disinfecting patient's unit by using VYV led lights and QleanAir Scandinavia® air filtering device) in reducing the rate of new carriage acquisitions of MDROs (MRSA, VRE, CRE, A. baumannii, P. aeruginosa, C. difficile).
   2. Analyze the role of a comprehensive intervention (consisting of establishing a "patient's unit commando" team, while continuously disinfecting patient's unit by using VYV led lights and QleanAir Scandinavia® air filtering device) in reducing the incidence of HA-BSI.
   3. Analyze the role of a comprehensive intervention (consisting of establishing a "patient's unit commando" team, while continuously disinfecting patient's unit by using VYV led lights and QleanAir Scandinavia® air filtering device) in reducing the incidence of HAUTI.

      Study protocol
      1. Prospective cluster-randomized placebo-controlled cross-over study design.
      2. The study will be conducted over 15 months; each study phase will last 6 months, with a pre-study period (1 month), a washout period (1 month) and a post study period (1 month).

         • Pre-study period: all patient rooms at both departments will be cleaned and disinfected according to the "common practice" as detailed below.

         • Phase I:

         o Medicine A: cleaning of patients' rooms will be subjected to a comprehensive intervention, consisting of: 1) a "patient's unit commando" team for daily and for terminal cleaning, 2) all lights in patients' room are VYV led lights, and 3) in each room, a QleanAir Scandinavia® filtering machine will be placed.
         * Medicine B: patients' rooms will be cleaned and disinfected according to the current "common practice" as detailed below.

           • Washout period in both hospitals: all patient rooms at both departments will be cleaned and disinfected according to the "common practice" as detailed below.

           • Phase II:
         * Medicine A: patients' rooms will be cleaned and disinfected according to the current "common practice" as detailed below.
         * Medicine B: cleaning of patients' rooms will be subjected to a comprehensive intervention, consisting of: 1) a "patient's unit commando" team for daily and for terminal cleaning, 2) all lights in patients' room are VYV led lights, and 3) in each room, a QleanAir Scandinavia® filtering machine will be placed.

           * Post-study period: all patient rooms at both departments will be cleaned and disinfected according to the "common practice" as detailed below.
           * The "patient's unit commando" team will consist of 6 staff members, trained specifically by the infection control team at Shamir Medical Center. The "patient's unit commando" team will be responsible, during the intervention, for the daily cleaning of the patients subjected to isolation precautions, and will be conducting the terminal cleaning following discharge of every patient from the unit that is under the intervention.

         Microbiological studies:

         • Clinical cultures are all processed at the SMC clinical microbiology laboratory. The laboratory adhere to the U.S. Clinical Laboratory Standards Institute (CLSI) standards and criteria. No additional cultures will be obtained specifically for this protocol.

         o MRSA, VRE, A. baumannii, and P. aeruginosa will be determined according to a Vitek-2 automated system and according to CLSI breakpoints and criteria.

         o CRE will be determined according to the Israeli MOH national diagnostic guidelines (2013) and based, again, on CLSI criteria.

         o Toxin-producing C. difficile will be determined based of a GDH-based serology test (C. DIFF QUIK CHEK COMPLETE®; Alere™) and if necessary (i.e., inconclusive serology test result: positive for C. difficile GDH antigen but negative for C. difficile toxins), will be confirmed by a PCR-based test (Xpert® C. difficile; Cepheid©). Samples will be processed according to national Israeli guidelines (2013) and according to CLSI criteria.

         o All MDROs will be stored in -800C for future molecular analyses.

         • Representative MDROs will be typed later on for future detailed transmission dynamics investigations.
         * The laboratory will be blinded to the source of the cultures (i.e., to the fact of whether or not the unit is at its interventional phase).

         Patients:

1. The two departments will perform, per local Infection Control regulations: i. Nasal culture for MRSA upon admission to the unit and weekly thereafter (same day and shift every week).

ii. Rectal culture for VRE, and CRE upon admission to the unit and weekly thereafter (same day and shift every week).

iii. Sputum and skin cultures (using sponges) for the presence of A. baumannii and P. aeruginosa upon admission to the unit and weekly thereafter (same day and shift every week).

2. All the surveillance for MDRO new acquisitions and hospital-acquired bloodstream infections (BSI) are conducted routinely and continuously by the Infection Control team at SMC. The PI serves as the head of the Infection Control unit and is personally involved in the surveillances processes for those endpoints.

3. Acquisitions of pre-specified MDROs:

1. MDRO acquisition will be defined based on clinical samples obtained from previously-not-known carriers. In addition, surveillance cultures for all the MDRO of interest (except C. difficile) would be obtained upon admission and weekly thereafter. An acquisition will be defined as a patient who was negative upon admission but became positive ≥ 72 hours after admission or within 72 hours after admission if the patient was hospitalized in the hospital during the last 30 days.
2. MRSA, VRE, and P. aeruginosa will be determined according to the Vitek-2 automated system and according to Clinical and Laboratory Standards Institute (CLSI) criteria.
3. CRE will be determined according to the Israeli ministry of health (MOH) national diagnostic guidelines (2013) and based, again, of the CLSI cutoffs and criteria.
4. C. difficile infection will be determined according to the Israeli ministry of health (MOH) national guidelines (2012), based on the presence of toxin-producing organism: first by GDH-based serology test and if needed, by confirmatory PCR-based test.
5. The monitoring and surveillance of hospital-acquired BSI, conducted by Infection Control personnel, is based on the Israeli Ministry of Health monitoring criteria, which resembles exactly the U.S. Centers for disease Control and Prevention (CDC) criteria.
6. The monitoring and surveillance of hospital-acquired UTI, conducted by Infection Control personnel, is based on the Israeli Ministry of Health monitoring criteria from 2014, which resembles (but is not exactly the same) as the U.S. CDC diagnostic criteria.

Power calculations

The power calculations are based on the primary study outcome, which is the MDRO new acquisitions incidence. Based on surveillance data from SMC, during 2019, the incidence (in the two departments) of MDRO new acquisition was 4.1 per 1,000 patient days. Even if the impact of the intervention would be relatively mild, and it will reduce the acquisition rate by only 10%, the sample size will still enable us with β=0.8 and α=0.01 to determine the statistical significant efficacy of the intervention.

Statistical analysis

Data will be summarized with descripted statistic based on the Data reference sheet.

The two groups (department ) will be compared for admission data, baseline characteristics and risk factors with the independent t-test and the Chi-Square test. . New carriage acquisitions of MDROs (MRSA, VRE, CRE, A. baumannii, P. aeruginosa, C. difficile), the incidence of HA-BSI and incidence of HAUTI will point estimated by rates, followed by 95% confidence interval.

Each department will be test for difference between the control and treatment period by the McNemar test for paired proportions.

Comparisons between study groups will be made by Z test for proportions for each Phase separately and for the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at Medicine A or Medicine B, Shamir (Assaf Harofeh) Medical Center.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-02-02 (Estimated); Study Completion 2025-08-03 (Estimated)

PRIMARY OUTCOMES:
Acquisitions of pre-specified MDROs: | 6 months
  Incidence of MDRO new carriage acquisitions (per 1,000 patient-days).

SECONDARY OUTCOMES:
Acquisitions of hospital acquired bloodstream infection | 6 months
  The hospital acquired bloodstream infection (HA-BSI) incidence (per 1,000 patient-days).
Acquisitions of ospital acquired urinary-tract infection (HAUTI) incidence (per 1,000 patient-days). | 6 months
  The hospital acquired urinary-tract infection (HAUTI) incidence (per 1,000 patient-days).

CONTACTS AND LOCATIONS:
Overall Officials: Dror Marchaim, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Shamir Medical Center (Assaf Harofeh), Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turner RM, White IR, Croudace T; PIP Study Group. Analysis of cluster randomized cross-over trial data: a comparison of methods. Stat Med. 2007 Jan 30;26(2):274-89. doi: 10.1002/sim.2537. PMID 16538700
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699
- [Background] Han JH, Sullivan N, Leas BF, Pegues DA, Kaczmarek JL, Umscheid CA. Cleaning Hospital Room Surfaces to Prevent Health Care-Associated Infections: A Technical Brief. Ann Intern Med. 2015 Oct 20;163(8):598-607. doi: 10.7326/M15-1192. Epub 2015 Aug 11. PMID 26258903
- [Background] Tanner WD, Leecaster MK, Zhang Y, Stratford KM, Mayer J, Visnovsky LD, Alhmidi H, Cadnum JL, Jencson AL, Koganti S, Bennett CP, Donskey CJ, Noble-Wang J, Reddy SC, Rose LJ, Watson L, Ide E, Wipperfurth T, Safdar N, Arasim M, Macke C, Roman P, Krein SL, Loc-Carrillo C, Samore MH. Environmental Contamination of Contact Precaution and Non-Contact Precaution Patient Rooms in Six Acute Care Facilities. Clin Infect Dis. 2021 Jan 29;72(Suppl 1):S8-S16. doi: 10.1093/cid/ciaa1602. PMID 33512527
- [Background] Ashkenazi H, Malik Z, Harth Y, Nitzan Y. Eradication of Propionibacterium acnes by its endogenic porphyrins after illumination with high intensity blue light. FEMS Immunol Med Microbiol. 2003 Jan 21;35(1):17-24. doi: 10.1111/j.1574-695X.2003.tb00644.x. PMID 12589953
- [Background] Manoukian S, Stewart S, Graves N, Mason H, Robertson C, Kennedy S, Pan J, Haahr L, Dancer SJ, Cook B, Reilly J. Evaluating the post-discharge cost of healthcare-associated infection in NHS Scotland. J Hosp Infect. 2021 Aug;114:51-58. doi: 10.1016/j.jhin.2020.12.026. PMID 34301396
- [Background] Maclean M, MacGregor SJ, Anderson JG, Woolsey G. Inactivation of bacterial pathogens following exposure to light from a 405-nanometer light-emitting diode array. Appl Environ Microbiol. 2009 Apr;75(7):1932-7. doi: 10.1128/AEM.01892-08. Epub 2009 Feb 6. PMID 19201962
- [Background] Wolkewitz M, Barnett AG, Palomar Martinez M, Frank U, Schumacher M; IMPLEMENT Study Group. Interventions to control nosocomial infections: study designs and statistical issues. J Hosp Infect. 2014 Feb;86(2):77-82. doi: 10.1016/j.jhin.2013.09.015. Epub 2013 Oct 18. PMID 24286854
- [Background] Boyce JM. Modern technologies for improving cleaning and disinfection of environmental surfaces in hospitals. Antimicrob Resist Infect Control. 2016 Apr 11;5:10. doi: 10.1186/s13756-016-0111-x. eCollection 2016. PMID 27069623
- [Background] Weber DJ, Rutala WA, Miller MB, Huslage K, Sickbert-Bennett E. Role of hospital surfaces in the transmission of emerging health care-associated pathogens: norovirus, Clostridium difficile, and Acinetobacter species. Am J Infect Control. 2010 Jun;38(5 Suppl 1):S25-33. doi: 10.1016/j.ajic.2010.04.196. PMID 20569853
- [Background] McKenzie K, Maclean M, Grant MH, Ramakrishnan P, MacGregor SJ, Anderson JG. The effects of 405 nm light on bacterial membrane integrity determined by salt and bile tolerance assays, leakage of UV-absorbing material and SYTOX green labelling. Microbiology (Reading). 2016 Sep;162(9):1680-1688. doi: 10.1099/mic.0.000350. Epub 2016 Aug 5. PMID 27499074